CLINICAL TRIAL: NCT00857740
Title: Influence of Painphysiolgy Education on the Pain Inhibition in Fibromyalgia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Dra. Jessica Van Oosterwijck, Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BUN B14320084324
Record Dates: First submitted 2009-03-06; First posted 2009-03-09 (Estimated); Last update posted 2010-07-08 (Estimated); Status verified 2009-03

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

INTERVENTIONS:
Behavioral: Education — Education about the neurophysiology of pain

SUMMARY:
The purpose of this study is to investigate whether education about the neurophysiology of pain is able to improve central pain inhibition in patients with Fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnose fibromyalgia
* Widespread pain
* Dutch speaking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Diffuse noxious inhibitory control | baseline, 14 days and 3 months follow-up

SECONDARY OUTCOMES:
pain pressure thresholds | baseline, 14 days and 3 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Van Oosterwijck, Doctoranda, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- Vrije Universiteit Brussel, Brussels, Brussels Capital, Belgium